CLINICAL TRIAL: NCT06623305
Title: Photobiomodulation Therapy for the Prevention and Treatment of Mucositis in Pediatric Oncology Patients
Brief Title: A Clinical Trial of the Administration of Light Therapy to Prevent and Treat Mouth Sores in Children With Cancer
Acronym: PBM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Elissa Shulta, Principal Investigator, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00051962
Record Dates: First submitted 2024-09-27; First posted 2024-10-02 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Mucositis Oral
Keywords: Photobiomodulation; Mucositis; Oral Mucositis
MeSH Terms: conditions — Stomatitis; Mucositis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Prospective - Retrospective Longitudinal Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Retrospective Arm (No Intervention): Retrospective data review of patients who did not receive light therapy
- Prospective Arm (Active Comparator): Prospective data review of patients who receive light therapy
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Light therapy will be administered using the cluster probe on the external cheeks bilaterally and intraorally using the lollipop probe for patients ≥7 years of age. Patients < 7 years of age will not receive intraoral treatment with the lollipop. Instead, they will be asked to open their mouth while the covered cluster probe is held externally to treat their intraoral membranes. Each treatment (both external cheeks and intraoral buccal region) will be administered over 1 min with a Modulation Frequency 2.5Hz, Skin Conduction nS 001, and Beam Power mW 000, for a total treatment time of 3 minutes.
  Other Names: PBM
  Arms: Prospective Arm

SUMMARY:
The goal of this clinical trial is to learn if light therapy can prevent and/or treat mouth sores in children with cancer. The main questions it aims to answer are:

Is it reasonable and acceptable to provide light therapy for children with cancer?

Does light therapy prevent and treat mouth sores related to medical treatment?

Researchers will compare children who did not receive light therapy before the clinical trial to children who receive light therapy during the clinical trial to see if light therapy helps to prevent and treat mucositis.

Participants will:

* Tell the nurse their pain score, related to their mouth sores, before receiving light therapy.
* Have picture taken of their mouth to look for mouth sores.
* Receive light therapy every other day while admitted to the hospital on the cancer unit or while admitted to an alternate unit.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to oncology unit, PICU, or on an alternate acute care unit.
* Diagnosis:
* Following diagnoses until achieve count recover (ANC≥500), the patient has no clinical signs of mucositis, or is discharged i. ALL interim-maintenance high dose Methotrexate ii. ALL with trisomy 21 receiving high dose Methotrexate iii. AML iv. Neuroblastoma (excluding admissions for antibody treatment) v. Burkitt lymphoma vi. Osteosarcoma receiving high dose Methotrexate vii. Germ cell tumors receiving Etoposide viii. Rhabdomyosarcoma ix. Ewing sarcoma
* Head/neck cancers receiving radiation
* Able to speak and understand English or Spanish

Exclusion Criteria:

* Unwilling to participate
* Do not meet eligibility criteria outline above

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility and acceptability of using PBM in pediatric oncology patients. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed through a questionnaire completed by the RN administering the PBM therapy and will focus on the patient's tolerance level rated on a numerical scale, the nurse's perception of feasibility, and length of treatment in minutes.

SECONDARY OUTCOMES:
Evaluate the effectiveness of using PBM based on mucositis onset | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record based on the first day a patient has reported oral mucosal pain or oral ulcers/sloughing.
Evaluate the effectiveness of using PBM based on mucositis severity. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record, defined using the CTCAE oral mucositis grading scale.
Evaluate the effectiveness of using PBM based on mucositis duration. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record, defined as the first day a patient has reported oral mucosal pain or oral ulcers/sloughing until the patient no longer reports oral mucosal pain or no longer has clinical signs of mucositis.
Evaluate the effectiveness of using PBM based on length of stay. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record, defined as the period of time between the patient's admission date and their discharge date.
Evaluate the effectiveness of using PBM based on narcotic usage. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record, defined as any narcotic administration documented in the Medication Administration Record, such as PRN narcotics (PO or IV), scheduled narcotics, or use of Patient-Controlled Analgesic.
Evaluate the effectiveness of using PBM based on nutritional support. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record, defined as the administration of TPN or lipids as documented in the Medication Administration Record.
Evaluate the effectiveness of using PBM based on pain score. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record, defined as the numeral rating that patient provides to the PBM RN using an age-appropriate pain scale specifically related to oral or throat pain.
  * 0 - 10: Verbal Numeric Rating Scale (VNRS)- Use for children ≥8 years old who understand the concept of order and number
  * Bieri Faces- Use for children > 3 years old who can understand the scale
  * FLACC - Revised (Face- Legs- Activity- Cry- Consolability)- Use for infants, toddlers, children with developmental delay, or any child who is unable to use a self-report scale (0-10 or Bieri faces)
Evaluate the effectiveness of using PBM based on MBI CLABSI rate. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record, defined as the rate of MBI CLABSIs per 1,000 line days.
Evaluate the effectiveness of using PBM based on Glutamine administration. | From date of enrollment until date of last PBM treatment, assessed up to 2 years.
  This will be assessed by the study team through analysis of retrospective and prospective data entered into the electronic health record, defined as a documented administration as "given" in the Medication Administration Record for oral glutamine in the past 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zadik Y, Arany PR, Fregnani ER, Bossi P, Antunes HS, Bensadoun RJ, Gueiros LA, Majorana A, Nair RG, Ranna V, Tissing WJE, Vaddi A, Lubart R, Migliorati CA, Lalla RV, Cheng KKF, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of photobiomodulation for the management of oral mucositis in cancer patients and clinical practice guidelines. Support Care Cancer. 2019 Oct;27(10):3969-3983. doi: 10.1007/s00520-019-04890-2. Epub 2019 Jul 8. PMID 31286228
- [Background] Treister NS, London WB, Guo D, Malsch M, Verrill K, Brewer J, Margossian S, Duncan C. A Feasibility Study Evaluating Extraoral Photobiomodulation Therapy for Prevention of Mucositis in Pediatric Hematopoietic Cell Transplantation. Photomed Laser Surg. 2016 Apr;34(4):178-84. doi: 10.1089/pho.2015.4021. Epub 2016 Mar 16. PMID 26982624
- [Background] Miranda-Silva W, da Fonseca FP, Gomes AA, Mafra ABB, Rocha V, Fregnani ER. Oral mucositis in paediatric cancer patients undergoing allogeneic hematopoietic stem cell transplantation preventively treated with professional dental care and photobiomodulation: Incidence and risk factors. Int J Paediatr Dent. 2022 Mar;32(2):251-263. doi: 10.1111/ipd.12850. Epub 2021 Jul 20. PMID 34115428
- [Background] Lima AG, Antequera R, Peres MP, Snitcosky IM, Federico MH, Villar RC. Efficacy of low-level laser therapy and aluminum hydroxide in patients with chemotherapy and radiotherapy-induced oral mucositis. Braz Dent J. 2010;21(3):186-92. doi: 10.1590/s0103-64402010000300002. PMID 21203698
- [Background] Heimlich FV, de Arruda JAA, Pereira NM, Faria LDS, Abreu LG, Ferreira MVL, Kakehasi FM, Travassos DV, Silva TA, Mesquita RA. Proposal of a prophylactic photobiomodulation protocol for chemotherapy-induced oral and oropharyngeal mucositis: a randomized clinical trial. Lasers Med Sci. 2023 Oct 27;38(1):245. doi: 10.1007/s10103-023-03916-w. PMID 37889325
- [Background] Chaves ME, Araujo AR, Piancastelli AC, Pinotti M. Effects of low-power light therapy on wound healing: LASER x LED. An Bras Dermatol. 2014 Jul-Aug;89(4):616-23. doi: 10.1590/abd1806-4841.20142519. PMID 25054749
- [Background] Antunes HS, Herchenhorn D, Small IA, Araujo CMM, Viegas CMP, de Assis Ramos G, Dias FL, Ferreira CG. Long-term survival of a randomized phase III trial of head and neck cancer patients receiving concurrent chemoradiation therapy with or without low-level laser therapy (LLLT) to prevent oral mucositis. Oral Oncol. 2017 Aug;71:11-15. doi: 10.1016/j.oraloncology.2017.05.018. Epub 2017 Jun 3. PMID 28688677
- [Result] Cheng KK, Lee V, Li CH, Yuen HL, Epstein JB. Oral mucositis in pediatric and adolescent patients undergoing chemotherapy: the impact of symptoms on quality of life. Support Care Cancer. 2012 Oct;20(10):2335-42. doi: 10.1007/s00520-011-1343-1. Epub 2011 Dec 14. PMID 22167295
- [Result] Pritchard M, Ogg SW, Bosi J, Mandrell BN. Utilization of Photobiomodulation for the Prevention and Treatment of Oral Mucositis. J Pediatr Hematol Oncol Nurs. 2024 Mar-Apr;41(2):107-113. doi: 10.1177/27527530231214525. Epub 2024 Feb 20. PMID 38377968
- [Result] Hafner D, Hrast P, Tomazevic T, Jazbec J, Kavcic M. Photobiomodulation for Chemotherapy-Induced Oral Mucositis in Pediatric Patients. Biomolecules. 2023 Feb 23;13(3):418. doi: 10.3390/biom13030418. PMID 36979353
- [Result] de Farias Gabriel A, Silveira FM, Curra M, Schuch LF, Wagner VP, Martins MAT, da Silveira Matte U, Siebert M, Botton MR, Brunetto AT, Gregianin LJ, Martins MD. Risk factors associated with the development of oral mucositis in pediatric oncology patients: Systematic review and meta-analysis. Oral Dis. 2022 May;28(4):1068-1084. doi: 10.1111/odi.13863. Epub 2021 Apr 9. PMID 33774891
- [Result] Berger K, Schopohl D, Bollig A, Strobach D, Rieger C, Rublee D, Ostermann H. Burden of Oral Mucositis: A Systematic Review and Implications for Future Research. Oncol Res Treat. 2018;41(6):399-405. doi: 10.1159/000487085. Epub 2018 May 3. PMID 29734184
- [Result] Antunes HS, de Azevedo AM, da Silva Bouzas LF, Adao CA, Pinheiro CT, Mayhe R, Pinheiro LH, Azevedo R, D'Aiuto de Matos V, Rodrigues PC, Small IA, Zangaro RA, Ferreira CG. Low-power laser in the prevention of induced oral mucositis in bone marrow transplantation patients: a randomized trial. Blood. 2007 Mar 1;109(5):2250-5. doi: 10.1182/blood-2006-07-035022. Epub 2006 Oct 19. PMID 17053058
- [Result] Alsheyyab F, Al-Momani D, Kasht R, Kamal A, Abusalem D, Al-Qasem W. Impact of severe oral mucositis in pediatric cancer patients on resource utilization and cancer treatment plans. Int J Clin Pharm. 2021 Oct;43(5):1322-1326. doi: 10.1007/s11096-021-01253-y. Epub 2021 Mar 3. PMID 33660192